CLINICAL TRIAL: NCT05471895
Title: Impact Des Violences Sexuelles Sur l'Incidence Des Interruptions Volontaires de Grossesses à La Réunion/ Impact of Sexual Violence on the Incidence of Voluntary Termination of Pregnancy in La Réunion
Brief Title: Impact of Sexual Violence on the Incidence of Voluntary Termination of Pregnancy in La Réunion
Acronym: IVIIRun
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/CHU/28
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-07

CONDITIONS: Sexual Violence; Abortion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to the figures for the last three years collected from the Indian Ocean Regional Health Observatory, it appears to be about twice as many voluntary terminations of pregnancy on the island of Reunion compared with France metropolitain region.

Furthermore, the overseas section in 2002, which looked at violence against women of all types in three different spheres of life (the marital sphere, the workplace and public spaces), tends to show a much higher incidence of sexual violence than in metropolitain France.

This trend seems to be confirmed by the overseas section of the VIRAGE survey started in 2018 on the island.

Furthermore, data found in a qualitative study conducted in Ile de France in 2013 seems to demonstrate a more frequent use of abortion among patients who are victims of sexual violence.

Thus, thiçs study will consist in evaluating the impact of sexual violence on the incidence of voluntary termination of pregnancy in Reunion Island.

ELIGIBILITY:
Inclusion Criteria:

- Adult patient coming for an abortion request at the CHU SUD and NORD, at the GHER and at the CEPS for the CHOR (Reunion Island)

Exclusion Criteria:

* Patient coming to the above-mentioned centres for a "post-abortion" consultation.
* <18 years
* Patient who does not speak French.
* Illiterate patient.
* Patient who has already completed the questionnaire.
* Patient refusing to participate in the study.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Each centre receives an average of 15 patients per day for pre-abortion consultations.
  Expectation of 7 fully completed questionnaires per day per centre, then approximately 1000 fully completed questionnaires for a total of 8 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of women victims of sexual abuse coming for a voluntary termination of pregnancy | Day 1
  Number of patients coming for a voluntary termination of pregnancy sexually abused

CONTACTS AND LOCATIONS:
Overall Officials: Véronique PERETTI, MD, Principal Investigator — CHU La Réunion

IPD SHARING:
Plan to Share IPD: No